CLINICAL TRIAL: NCT04660240
Title: Randomized Trial Investigating Clinical Outcomes of Two Sirolimus-Eluting Stents in Diabetes Mellitus
Brief Title: Randomized Trial Comparing Two Sirolimus-Eluting Stents in Diabetes Mellitus
Acronym: INC-DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Julio Ivan Farjat Pasos, Co-Principal Investigator, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INCAR-DG-DI-342-2020
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus; Coronary Artery Disease; Acute Coronary Syndrome
Keywords: Diabetes Mellitus; Albuminus; Orsiro; Percutaneous coronary intervention
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Diabetic patients undergoing percutaneous coronary intervention in de novo lesions are going to be randomized to two groups. One will have percutaneous coronary intervention with Abluminus sirolimus eluting stent implantation, and the other will have percutaneous coronary intervention with Orsiro Sirolimus Eluting stent implantation. The implantation of both stents will be guided by angiography only. In a subgroup of both arms (100 patients per group) the implantation will be also guided by intravascular ultrasound.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abluminus Sirolimus Eluting Stent System (ASES) (Active Comparator): The Abluminus sirolimus eluting stent manufactured by Envision and distributed by Concept Medical.
  Interventions: Device: Abluminus Sirolimus Eluting Stent System (ASES)
- Orsiro Sirolimus Eluting Coronary Stent System (OSES) (Experimental): The Orsiro sirolimus eluting stent manufactured by Biotronik.
  Interventions: Device: Orsiro Sirolimus Eluting Coronary Stent System (OSES)

INTERVENTIONS:
Device: Abluminus Sirolimus Eluting Stent System (ASES) — The procedure will be conducted in accordance with the CE mark instructions for use for the ASES.
  The need or not for postdilation in any segment of the stent will be at the discretion of the operator, seeking its adequate expansion and apposition. To consider PCI to be successful, residual stenosis must be less than or equal to 30% by angiography at the end of the procedure, including the absence of coronary dissection that compromises distal flow or a hemodynamically significant pressure gradient across the lesion.
  Arms: Abluminus Sirolimus Eluting Stent System (ASES)
Device: Orsiro Sirolimus Eluting Coronary Stent System (OSES) — The procedure will be conducted in accordance with the CE mark instructions for use for the OSES.
  The need or not for postdilation in any segment of the stent will be at the discretion of the operator, seeking its adequate expansion and apposition. To consider PCI to be successful, residual stenosis must be less than or equal to 30% by angiography at the end of the procedure, including the absence of coronary dissection that compromises distal flow or a hemodynamically significant pressure gradient across the lesion.
  Arms: Orsiro Sirolimus Eluting Coronary Stent System (OSES)

SUMMARY:
Randomized, controlled, blind, single-center and non-inferiority clinical trial to compare the target lesion failure (TLF) at 12 months in patients with diabetes mellitus who underwent percutaneous coronary intervention with an Orsiro stent vs. Abluminus stent.

DETAILED DESCRIPTION:
Worldwide, and especially in Mexico, there is a high incidence of diabetes mellitus (DM), which in turn, confers a higher cardiovascular risk in this population. Diabetic patients undergoing PCI have worse outcomes than non-diabetics regardless of the degree of complexity of their coronary anatomy. Although the 30-day in-hospital outcomes have been similar between diabetic and non-diabetic patients, DM has been invariably associated with greater stent failure with target vessel revascularization (TVR), major adverse cardiovascular event (MACE), and mortality in the long-term follow-up, even with the use of drug-eluting stents. In relation to the above, two of the sirolimus-eluting stents (SES): the Abluminus and the Orsiro, have been considered as promising options in patients with DM. The Abluminus stent has been designed for diabetic patients in order to reduce cardiovascular events. Said stent consists of a cobalt-chromium platform covered with a layer of biodegradable polymer and mounted on a balloon, both sirolimus-releasing. The Rate of target lesion failure (TLF) reported to date in diabetic patients is 3.8%. On the other hand, the Orsiro stent, a cobalt-chromium platform with ultrathin struts, has had favorable results in different clinical settings and patients with different characteristics]; specifically in a subgroup analysis in DM, a TLF rate of 3.5% was reported

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age.
* Provide informed consent and agree to follow up as stipulated in the protocol.
* Diabetes mellitus. Whether it is DM 1 or 2 previously diagnosed or newly diagnosed by:

  * Fasting glucose> 126 mg / dl (for study terms, fasting will be defined as the absence of caloric intake for> 8 hours)
  * Tolerance curve to glucose (75 grams of glucose orally) with a glycemia at 2 hours> 200 mg / dl or,
  * HbA1C> 6.5%.
* Coronary artery disease including chronic coronary syndrome, silent ischemia, or non-ST-segment elevation acute coronary ischemic syndrome.
* Presence of 1 or more de novo coronary lesions in native coronary arteries with a site of maximum stenosis> 50% that may be amenable to stenting; without limitation in the number of lesions or vessels affected.

Exclusion Criteria:

* Cardiogenic shock.
* Allergy to acetylsalicylic acid, clopidogrel, ticagrelor, prasugrel, heparin, sirolimus or contrast medium, which cannot be adequately premedicated.
* Acute ST-segment elevation myocardial infarction candidate for primary or urgent coronary angioplasty.
* Left main coronary artery disease.
* In-stent restenosis.
* Lesions in venous or arterial grafts.
* Surgery (cardiac or non-cardiac) planned within 6 months of PCI, unless dual antiplatelet therapy can be continued in the periprocedural period.
* Inability to provide informed consent.
* Life expectancy <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Target Lesion Failure (TLF) | 12 months
  To compare the rate of target lesion failure (composed of cardiovascular death, myocardial infarction related to the treated vessel or ischemia driven target lesion revascularization)

SECONDARY OUTCOMES:
Cardiovascular Death | 12 months
  Cardiovascular death is defined as death resulting from cardiovascular causes. The following categories may be collected:
  * Death caused by acute MI
  * Death caused by sudden cardiac, including unwitnessed, death
  * Death resulting from heart failure
  * Death caused by stroke
  * Death caused by cardiovascular procedures
  * Death resulting from cardiovascular hemorrhage
  * Death resulting from other cardiovascular cause
    * Any MI not clearly attributable to a non-target vessel will be considered as target-vessel MI.
    * Percutaneous coronary intervention (PCI) related MI is termed type 4a MI.
    * Coronary artery bypass grafting (CABG) related MI is termed type 5 MI. Revascularization is clinically driven if the target lesion diameter stenosis is > 50% by quantitative coronary angiography (QCA) and the subject has clinical or functional ischemia which cannot be explained by another native coronary or bypass graft lesion.
Myocardial Infarction (MI) | 12 months
  Compare the myocardial infarction related to the treated vessel between both groups.
  (according to the 4th international definition of myocardial infarction) detection of an increase or decrease in cardiac troponin values with at least 1 of the values above the upper reference limit of the 99th percentile and at least 1 of the following conditions :
  * Symptoms of acute myocardial ischemia.
  * New ischemic changes in the electrocardiogram.
  * Appearance of pathological Q waves.
  * Imaging evidence of loss of viable myocardium or new regional abnormalities in myocardial wall mobility following a pattern compatible with ischemic etiology.
  * Identification of a coronary thrombus by angiography with intracoronary imaging or by autopsy
    * Any MI that cannot be clearly attributed to a vessel other than the revascularized one will be considered as MI related to the treated vessel.
Target Lesion Revascularization (TLR) | 12 months
  Revascularization is clinically driven if the target lesion diameter stenosis is > 50% by quantitative coronary angiography (QCA) and the subject has clinical or functional ischemia which cannot be explained by another native coronary or bypass graft lesion.
Target vessel revascularization (TVR) | 12 months
  TVR is a repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.
Target vessel failure (TVF) | 12 months
  To compare the rate of target vessel failure (composed of cardiovascular death, myocardial infarction related to the treated vessel or ischemia driven target vessel revascularization)
Death caused by other cardiovascular causes. | 12 months
  Compare death from any cause between the two groups.
  The following categories will be collected:
  * Malignancy.
  * Pulmonary causes.
  * Infection.
  * Gastrointestinal causes.
  * Accident / trauma.
  * Caused by failure of another non-cardiovascular organ.
  * Other non-cardiovascular causes.
    * Death that cannot be attributed to any of the aforementioned categories due to lack of information will be considered cardiovascular in terms of study outcomes.
Rate of in-stent restenosis (ISR) | 12 months
  Compare the rate of stent edge restenosis between both groups. Stenosis> 50% of the diameter and one or more of the following: symptoms suggestive of ischemia, electrocardiographic changes suggestive of ischemia, significant pressure gradient across the lesion; or a> 70% reduction in luminal area, even in the absence of data suggestive of ischemia.
  The categories will be collected according to the Waksman In-Stent Restenosis Classification:
  * Type I: mechanical
    * IA Underexpansion
    * IIA Stent fracture
  * Type II: Biologic
    * IIA Intimal hyperplasia
    * IIB Neoatherosclerosis, noncalcified
    * IIC Neoatherosclerosis, calcified
  * Type III: Mixed pattern: Combined mechanical and biologic etiology
  * Type IV: Chronic total occlusion
  * Type V: >2 layers of stent
Rate of stent thrombosis (ST) | 12 months
  Compare the rate of stent thrombosis between both groups, According to the definition of the Academic Research Consortium (ARC) -2:
  1. Definitive thrombosis.
  2. Probable thrombosis.
  3. Silent occlusion.
  4. Temporality: acute (0-24 hours), subacute (> 24 hours to 30 days), late (> 30 days to 1 year) and very late (> 1 year).
Major bleeding | 12 months
  Compare the incidence of bleeding complications according to The Bleeding Academic Research Consortium 2 (BARC-2) scale: 3 or greater.
Rate of Cerebrovascular Event | 12 months
  Compare the rate of cerebrovascular event between both groups according to Neuro-ARC stroke/ Transient ischemic attack (TIA) criteria.
Contrast Nephropathy | 48 hours
  Creatinine increase >0.5 mg / dl or >25% over baseline at 48 hours after the procedure.
Technical Success | 12 months
  Technical success is defined as the ability to cross the occluded segment with both a wire and a balloon, and successfully open the artery; the restoration of antegrade Thrombolysis In Myocardial Infarction (TIMI) flow 2 or 3 and a <30% residual stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Guering Eid Lidt, MD, Study Director — Instituto Nacional de Cardiología Ignacio Chávez; Julio I Farjat Pasos, MD MSc, Principal Investigator — Instituto Nacional de Cardiología Ignacio Chávez; Walter O Magaña Ornelas, MD, Principal Investigator — Instituto Nacional de Cardiología Ignacio Chávez; Alejandra D Portillo Romero, MD, Principal Investigator — Instituto Nacional de Cardiología Ignacio Chávez; José A Ayón Martínez, MD, Principal Investigator — Instituto Nacional de Cardiología Ignacio Chávez
Locations (1):
- Instituto Nacional de Cardiología Ignacio Chávez, Mexico City, Tlalpan, Mexico